CLINICAL TRIAL: NCT02855554
Title: Novel Magnetic Resonance Imaging Techniques for Quantitative Cardiac Parametric Mapping
Brief Title: Quantitative Cardiac Parametric Mapping
Acronym: Myomapping
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00035552
Record Dates: First submitted 2016-07-28; First posted 2016-08-04 (Estimated); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Cardiomyopathy, Myocarditis, Ischemic Heart Disease
Keywords: myocardial tissue characterization
MeSH Terms: conditions — Cardiomyopathies; Myocarditis; Myocardial Ischemia | interventions — X-Rays

ARMS (1):
- Additional 5 minute research MR scan of heart. (Experimental): The purpose of this is to evaluate new, faster MR scans
  Interventions: Other: Cardiac Magnetic Resonance (CMR) imaging techniques

INTERVENTIONS:
Other: Cardiac Magnetic Resonance (CMR) imaging techniques — Evaluation of clinical potential of fast quantitative myocardial tissue characterization using recently emerged CMRI techniques to aid the diagnosis, treatment, and follow up of patients with myocardial diseases.

SUMMARY:
The overall goal of this project is to evaluate the clinical potential of fast quantitative myocardial tissue characterization using recently emerged Cardiac Magnetic Resonance Imaging (CMR) techniques to aid the diagnosis, treatment, and follow up of patients with myocardial diseases, such as ischemic heart disease, cardiomyopathies, and myocarditis.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18-90 years of age.
* Subject must be previously diagnosed with or suspected to have one of the following conditions.
* Myocardial ischemia or infarction (group 1)
* Hypertrophic cardiomyopathy (group 2)
* Infiltrative cardiomyopathy (group 3)
* Myocarditis (group 4)
* Subject must have been referred for a clinically indicated CMR.

Exclusion Criteria:

* Subject has any implanted device or condition in which an MR scan would be contraindicated.
* Subject has an acute psychiatric disorder or is cognitively impaired.
* Subject is using or is dependent on substances of abuse.
* Subject is unwilling to comply with the requirements of the protocol.
* Subject has previously entered this study.
* Subject has an allergy against MRI contrast agents.
* Subject is in acute unstable condition.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2014-06-20; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Clinical value of fast T1, T2, and T2* mapping of the left ventricle for the assessment of necrosis/scar, edema, and possible intramyocardial hemorrhage in patients with heart disease. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Akos Varga-Szemes, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States